CLINICAL TRIAL: NCT01219465
Title: Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cells Infusion for Initial Type 1 Diabetes
Brief Title: Umbilical Cord Mesenchymal Stem Cells Infusion for Initial Type 1 Diabetes Mellitus
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qingdao University (Other)
Responsible Party: Wang, Yangang MD, Stem Cell Research Center of Medical School Hospital of Qingdao University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSCT1DM003
Record Dates: First submitted 2010-10-12; First posted 2010-10-13 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-09

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Mesenchymal Stem Cells; Umbilical Cord
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; mesenchymal stem cells; Umbilical cord
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord mesenchymal stem cells (Experimental): Intravenous infusion of ex vivo cultured umbilical cord mesenchymal stem cells
  Interventions: Biological: umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: umbilical cord mesenchymal stem cells — Transfusion of the umbilical cord mesenchymal stem cells (2 x 107 cells) intravenously.
  Other Names: mesenchymal stem cells

SUMMARY:
The purpose of this study is to determine whether umbilical cord Mesenchymal Stem Cells of treatment for initial type 1 diabetes is safe and effective.

DETAILED DESCRIPTION:
Type 1 diabetes mellitus (T1DM)is characterized by the autoimmune destruction of the pancreatic β cells.Patients require multiple daily insulin injections throughout their lives as well as close monitoring of their diet and blood sugar levels to prevent complications. The investigators hope umbilical cord Mesenchymal Stem Cells could not only address the need for β-cell replacement but also control of the autoimmune response to β cells.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 1 diabetes by ADA criteria less than 9 weeks.
* Ability to provide written informed consent from patients or Child guardian.

Exclusion Criteria:

* diabetic ketoacidosis.
* evidence of retinopathy at baseline.
* Body Mass Index >30.
* Severe or acute organ damage.
* Infectious diseases, e.g. HIV infection, or hepatitis B or C infection.
* Severe psychiatric disorder.
* Presence of malignancy.

Ages: 3 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
C peptide release test | 3 months

SECONDARY OUTCOMES:
Exogenous insulin dose | 3 months
blood glucose | 3 months
glycosylated Hemoglobin A1c | 3 months
Number of severe and documented hypoglycemic events | 3 months
Immunologic reconstitution parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yangang Wang, MD Phd, Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- Stem Cell Research Center of Medical School Hospital of Qingdao University, Qingdao, Shandong, China